CLINICAL TRIAL: NCT00502684
Title: Perioperative Administration of COX 2 Inhibitors and Beta Blockers in Women Undergoing Breast Cancer Surgery: an Intervention to Decrease Immune Suppression, Metastatic Potential and Cancer Recurrence
Brief Title: Perioperative Administration of COX 2 Inhibitors and Beta Blockers to Women Undergoing Breast Cancer Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kaplan Medical Center (Other)
Collaborators: Tel Aviv University (Other); Tel-Aviv Sourasky Medical Center (Other Government); Sheba Medical Center (Other Government); Rabin Medical Center (Other)
Responsible Party: Principal Investigator, Tanir M Allweis, MD, Director, Sarah Markowitz Breast Health Center, Kaplan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 392-22.6.07 / 2358 HMO-CTIL
Record Dates: First submitted 2007-07-17; First posted 2007-07-18 (Estimated); Last update posted 2014-07-01 (Estimated); Status verified 2014-06

CONDITIONS: Primary Operable Breast Cancer
Keywords: breast cancer; surgery; immune suppression; beta blockers; COX2 inhibitors
MeSH Terms: conditions — Breast Neoplasms | interventions — Propranolol; Etodolac

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Peri-operative etodolac and propranolol as described in protocol
  Interventions: Drug: Propranolol, etodolac
- 2 (Placebo Comparator): peri-operative placebo as described in protocol

INTERVENTIONS:
Drug: Propranolol, etodolac — propranolol 10 mg X 4 /day, starting on day -3 pre-op, for 6 days, till POD 2 Etodolac 400 mg X2/day, starting on day -3 pre-op, for 6 days, till POD 2
  Arms: 1

SUMMARY:
Surgery for breast cancer has a major role in enhancing long term survival and cure, but several physiological aspects associated with surgery are implicated as enhancing tumor spread and formation of distant metastases. These include: an increase in pro-angiogenic factors, direct spread of tumor cells, accumulation of grown factors, immune suppression and direct effects of anesthetics and opiate pain relievers on cancer cells. Some of these pro-metastatic mechanism may be blocked by the interventions proposed in this study, namely by administration of beta-adrenergic blockers and COX2 inhibitors around the time of surgery.

Studies have shown that surgery increases levels of catecholamines and prostaglandins, which in turn may promote the release of pro-angiogenic factors such as VEGF, and enhance vascularization of micro metastases.

Opiates given for pain relief during and after surgery have been reported to enhance tumor cell division and cause immune suppression.

The immune system is significantly suppressed during surgery. This suppression has been shown to affect the systemic resistance to infection as well as neoplastic metastatic processes.

Several studies have shown that increased levels of catecholamines and prostaglandins add to the immune suppression.

Studies in rats found that peri-operative administration of the beta beta-blocker propranolol together with the COX2 inhibitor etodolac significantly reduced the suppression of NK cell activity as well as the risk for distant metastases.

A recent retrospective clinical study found that among breast cancer patients treated with a combination of regional anesthesia and a COX inhibitor the recurrence rated were significantly less than among patients undergoing surgery without these two interventions.

The purpose of the proposed prospective trial is to examine if peri-operative administration of the combination of a beta-blocker together with a COX2 inhibitor will prevent suppression of cellular immunity, decrease VEGF levels, and decrease cancer recurrence rates.

In the proposed study breast cancer patients will be treated with a combination of a beta-blocker and COX2 inhibitor (or placebo) before, during and after surgery. (A control group of healthy women will serve as untreated controls). The variables which will be examined are: number and activity of NK cells, levels of Th1 and Th2 cytokines, serum stress hormones and angiogenic factors, and the ability of leukocytes to produce Th1 and Th2 cytokines as a result of in vitro stimulation.

In addition to these immediate parameters, long term follow up will be conducted in order to determine the effect of the intervention on long term cancer recurrence over five years.

Statistical analysis will be done using t-tests, ANOVA, and multivariate regressions, with regard to the known risk factors for recurrence such as tumor grade, lymph node involvement etc. Sample size for immunological parameters will be 40 patients in each group and 20 healthy women. Sample size for estimates of cancer recurrence at five years of follow up wiil be 460 women (230 in each group). This sample size provides a power of 80% to detect a 50% reduction in cancer recurrence at an α of 0.05.

DETAILED DESCRIPTION:
Scientific Background Anesthesia and surgery are stressful situations which cause neuro-endocrine, metabolic and neurological responses. Cancer surgery may cause a decrease in anti-angiogenic factors, and enable dissemination of tumor cells through manipulation of the tumor and it blood vessels, as well as local and systemic secretion of growth hormones, and immune suppression. The magnitude of the response depends on many factors, including the extent of tissue injury, technique of anesthesia and type of analgesia, transfusions, temperature changes, psychological stress and genetic factors (1-3). The tissue damage starts a cascade of local and systemic processes which include secretion of hormones and cytokines (1).

Post operatively, suppression of several immune functions occurs, and may last for weeks. The cellular immunity undergoes suppression, while the humoral immunity remains almost entirely intact (1). These changes in cell mediated immunity may impact systemic resistance to infection as well as metastatic processes. Specifically, NK cells have a pivotal role in defense from neoplastic processes. Studies have shown that high levels of activity of NK cells are associated with long term survival (1). Therefore, understanding of the processes which cause post-operative immune suppression, and prevention of such suppression, are of clinical significance.

Several substances which are secreted after surgery are thought to contribute to immune suppression in general and NK cell dysfunction in particular. These include prostaglandins, catecholamines, steroids and endorphins, have all been shown to suppress several immunological functions in vitro (1). Animal studies have shown that administration of prostaglandins and catecholamines to rats suppresses NK cell activity in vivo, in association with elevated susceptibility to metastases 4-6).

In rats undergoing a laparotomy, peri-operative administration of beta- adrenergic blockers together with COX-2 inhibitors significantly abrogated the NK cell suppression as well as the enhanced susceptibility to metastases after surgery (4,7).

The mechanism of effect of prostaglandins and catecholamines on NK cells has been elucidated (1): beta- adrenergic receptors and prostanoid receptors on the cell membrane cause elevated levels of intra-cellular cAMP when activated by their ligand, which in turn interferes with the NK cell cytotoxic activity against cancer cells or viral pathogens. Since the elevated intra-cellular levels of cAMP is caused by each type of receptor independently, blockade of only one of these pathways will enable an increase in intracellular cAMP levels via the other pathway, and have no effect of the suppression of cytotoxic activity. Therefore, simultaneous blockade of both pathways may be more effective. Research in rats directly supports this hypothesis (7).

Cells of the immune system express mostly beta-2 adrenergic receptors, and to a lesser degree beta-1 receptors (9, 10), so pharmacological blockade requires use of a non specific blocker which can block both types of receptors. The beta-antagonist propranolol was chosen for this experiment since it is a non specific beta-blocker, capable of blocking both types of receptors, as well as extensive clinical experience with this drug and the fact that it is a relatively safe drug. The COX-2 inhibitor chosen is Etodlac (Etopan), which has the advantage of being a selective COX-2 inhibitor,synthesized during injury and inflammation, with little effect on the COX-1 enzyme, which is associated with ongoing maintenance of tissues.

Anesthetics and opiate analgesics also cause NK cell suppression. Research in animals and in humans has shown that morphine and fentanyl cause suppression of NK cell activity, and enhance susceptibility to breast cancer metastases in rats (11,12). Lower doses of opiates in patients have been reported to decrease the immune suppression magnitude and duration (13). Therefore, peri-operative interventions which decrease the use of opiates (or their endogenous secretion) may be clinically important factors in cancer recurrence.

In addition to immune suppression, endogenous and exogenous opiates (endorphins morphine, fentanyl) have been implicated as promoting metastatic spread and neoplastic proliferation via other mechanisms:

* Catecholamines have been reported to increase VEGF secretion by human cancer cells, and enhance tumor cell invasion (14-16).
* Morphine causes increased proliferation of human tumor cells and enhances tumor vascularization (17)
* COX2 inhibitors enhance sensitivity of human tumor cells to induction of apoptosis, and decrease capillary density in cancer tissue (18, 19).

Therefore, minimization of peri-operative opiate use and prevention or blockade of prostaglandin and catecholamine effects may delay the metastatic process and the development of existing micro-metastases.

A retrospective clinical study published in 2006 indirectly supports the proposed study: In this study breast cancer patients were treated per-operatively with a COX inhibitor (diclofenac) along with local blockade of the sympathetic and pain pathways (paravertebral anesthesia). These treatments no doubt lowered the use of opiates during and after surgery. Among patients thus treated a three fold decrease in recurrence rates was found three years after surgery (21). Of note, this study quotes the previously mentioned study in rats (6,22) and involves the same interventions.

AIM The aim of the proposed study is to examine whether peri-operative administration of COX2 inhibitors with beta- adrenergic blockers decreases immune suppression during surgery, decreases stress hormone and pro-angiogenic factor secretion, and is associated with a decrease in cancer recurrence rates.

The peri-operative variables which will be examined will include number and activity of NK cells in the blood, levels of Th1 and Th2 cytokines, stress hormones and pro-angiogenic factors, and Th1 and 2 cytokine production by leukocytes in response to in vitro stimulation. As part of the clinical monitoring meticulous recording of type and doses of analgesics given post operatively, as well as post operative pain assessment (NAS VAS). In addition to these parameters, long term follow up will be conducted to determine long term effects of the intervention on cancer recurrence.

Peri-operative administration of COX inhibitors and beta- adrenergic blockers Routine pre medication before surgery generally includes anxiolytics such as benzodiazepines, drugs routinely taken by the patient, and additional drugs for specific indications. Preventive administration of beta- blockers and COX inhibitors are recommended in the literature pertaining to anesthesia and pain. Administration of beta- blockers has been shown to stabilize the cardio vascular system and decrease peri-operative ischemic events (23), while preventive administration of COX inhibitors decreases post operative pain (5). Post operative pain has significant immunological effects: it causes secretion of endogenous opiates, and is often treated with synthetic opiates such as morphine. The opiates cause a stress response, suppress immune functions and promote tumor growth and spread. Studies have shown that administration of COX inhibitors together with morphine caused a decrease in morphine requirements. Administration of COX inhibitors can help control pain by abrogation of prostaglandin mediated pain pathways while at the same time decreasing opiate requirements. An additional benefit of COX inhibitors is it's direct activity against tumor cells by enhancing apoptosis and decreasing tumor blood supply as reported in a recently published study (21). These studies indicate that peri-operative use of these drugs does not have any detrimental effects, is not associated with increased complication - and in fact may be beneficial.

Patients and Methods

Patients and treatments:

Immune system activity will be determined among 80 operated breast cancer patients, and 20 health women in the following groups:

* Treatment arm: 40 patients undergoing elective surgery for primary breast cancer will be treated orally according to the following protocol:

  * Propranolol (Deralin) - patients will receive a low dose of 40 mg/day (4X10mg) starting two days before surgery (immediately following the first blood draw) until the evening of surgery. The first dose will be given under supervision (described later). On the morning of surgery, a single tablet of propranolol XL 80mg will be administered together with other pre-medication drugs, and will be continued once daily for three days after surgery. Pulse and blood pressure will be monitored during the first day of treatment, during the day of surgery and on the following days until discharge from the hospital. If pulse decreases to <50/min or blood pressure decreases to <100 systolic - the dose will be halved.
  * Etodolac (Etopan) - patients will receive 400mg of etodolac XL twice a day starting two days before and continuing through two days after surgery.
* Control arm: Forty patients undergoing the same operations will be treated with placebo drugs on the same schedule.
* Healthy controls: a third control arm will include 20 healthy age-matched women presenting for routine breast exams and not undergoing surgery will undergo blood tests only.

Patients will be randomized to one of the two groups, and patient, physicians and laboratory personnel will be blinded to the patient's assignment.

Dependent variables to be tested:

1. Cytotoxic activity of NK cells against K562 target cells.
2. Blood leukocyte levels of NK cells, NKT cells, lymphocytes, monocytes and granulocytes as determined by FACS.
3. Serum levels of cytokines (Th1, Th2 and inflammatory): IFN-gamma, IL-2, IL-12, IL-4, IL-10 IL-10 and IL-6.
4. In vitro cytokine secretion by leukocytes stimulated by HPA and LPS. (IFN-gamma IL- 2, IL-12, IL-4, IL-10 IL-10 and IL-6.)
5. Stress hormones and angiogenic factors: levels of cortisol and VEGF.
6. Doses of anesthetics and analgesics used during and after surgery.
7. Cancer recurrence during 5 years (including site of recurrence). In addition to the aforementioned groups, another 190 patients will be recruited onto each group without examining immunological parameters, and will be followed only for cancer recurrence.

Eligibility criteria:

* Women that are scheduled to undergo surgery of a single, stage I-III, invasive ductal or lobular carcinoma tumor with curative intent
* No evidence of metastatic disease prior to surgery. Minimal workup would include chest XR, abdominal ultrasound and bone scan.
* Age between 20 and 70 year old.
* ASA score of 1-2
* The patient is able to understand the study objectives and procedures, able to comply with the protocol, and is capable to sign an informed consent.

Exclusion criteria:

* Patients with metastatic disease, known prior to surgery.
* Patients in whom surgical resection is planned without curative intent.
* Patients who have undergone neoadjuvant treatment.
* Patients with renal failure, measured by creatinine level >1.5
* Patients with significant heart failure (NYHA functional class 3 or higher)
* Patients with significant liver failure (known cirrhosis, Bilirubin level>2)
* Patients suffering from asthma
* Patients with known allergy to one or more of the study medications
* Patients with known allergy to any medication from the non-steroidal anti-inflammatory drug group.
* Patients with diabetes mellitus (type 1 or 2).
* Patients treated chronically with one or more of the study medications
* Patients treated chronically with any type of Beta adrenergic blocker.
* Patients treated chronically with any type of COX inhibitor.
* Patients with second or third degree AV block.
* Patients with sinus bradycardia (patients with heart rate of less than 50).
* Patients with sick sinus syndrome.
* Patients with current atrial fibrillation/flutter.
* Patients with Printzmetal's angina
* Patients with hypertension
* Patients with right sided heart failure owing to pulmonary hypertension.
* Patients with significant cardiomegaly
* Patients with (current) pheochromocytoma
* Patients with chronic Digoxin treatment
* Patients with active peptic disease
* Patients with peripheral vascular disease
* Patients with history or concomitant malignant disease of any type other than breast cancer.
* Patients who were treated with chemotherapy in the last 10 years for any reason besides neo-adjuvant therapy for breast cancer within the last six months.
* Pregnant woman.
* Patients currently participating in any other clinical trial

Procedure:

After obtaining Helsinki committee approval, eligible patients will receive explanations and be invited to participate in the study. Women who consent will sign the approved informed consent form.

Anesthesia procedure will include:

Standard monitoring including automated blood pressure, ECG, O2 saturation, levels of inhaled and exhaled gases Pre-medication: at anesthesiologists discretion Induction: at anesthesiologist's discretion Maintenance: at anesthesiologist's discretion (an effort will be made to minimize opiate use but without compromising on pain control).

Post operative pain management:

Patients will be given a choice of oral Paracetamol 1000 mg every 4 hours, oral Dipyrone 1000 mg every 4 hours, oral Tramadol solution 50 mg every 6 hours and combinations of the above. If needed - 5 mg of oral percocet/oxycodone syrup every 6 hours may be added. For patients who are unable to sustain oral intake, intravenous Tramal will be offered at a dose of 50-100 mg every 6 hours and if needed - morphine 0.1 mg/kg every 4 hours. This protocol is identical to the one currently used after this type of surgery.

Blood samples :

Blood samples will be obtained two days before surgery (prior to administration of study drugs or placebo), on the morning of and the morning following surgery. Blood samples will be drawn between 7:30 and 9:00 am, and will include 10 cc of peripheral blood, preferably from the ante-cubital vein.

Blood will be collected in vacuum tubes containing 30 units of heparin without preservatives, and will be transferred immediately to the neuro-immunology lab at Tel Aviv University. Laboratory evaluation of the samples will begin within 3 hours of blood drawing. The samples will be kept at room temperature.

The samples will be divided as follows:

NK cell activity testing - 2 ml FACS analysis of cells - 1 ml In vitro testing of cytokine response to LPS - 2 ml Cytokine, cortisol and VEGF levels - 5 ml (to be performed in batches at a later time - after separation of cells plasma will be kept at -80C).

Documentation and analysis of results:

Documentation:

Epidemiological data: identification (name, ID no), age, ethnic origin, background medical conditions and drugs, smoking, menstrual status and date of last menstrual period, physical activity, presence of infections or viral illnesses within last 2 weeks.

Data related to anesthesia and surgery:

Type and length of surgery, systemic administration of opioids during and after surgery (type and dose).

Cancer related parameters: Tumor size, grade, histological type, lymph node status, adjuvant therapy.

Immunological parameters: as previously detailed is three blood samples from operated patients and a single sample from the healthy controls.

Recurrence data: location, time since surgery and survival.

Statistical Analysis:

Statistical analysis will be done by ANOVA (between and within subjects) regarding the variables. Determination of specific differences between groups will be based on the PLSD test for planned comparisons, and the Scheffe test for unplanned comparisons. Chi square tests will be used as well as Kaplan-Meier survival curves for non continuous or categorical variables. In addition, Cox regressions will be calculated to evaluate the predictive ability of treatments on cancer recurrence, taking other predicting factors into account. Blood samples and immunological data will be collected for 40 patients in groups 1 and 2 and 20 healthy controls in group 3. In order to determine impact of treatment on recurrence rates a total of 230 patients will be recruited in each group. Sample size was calculated to provide an 805 power to detect a 30-50% decrease in cancer recurrence with an alpha of 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Women that are scheduled to undergo surgery of a single, stage I-III, invasive ductal or lobular carcinoma tumor with curative intent
* No evidence of metastatic disease prior to surgery. Minimal workup would include chest XR, abdominal ultrasound and bone scan.
* Age between 20 and 70 year old.
* ASA score of 1-2
* The patient is able to understand the study objectives and procedures, able to comply with the protocol, and is capable to sign an informed consent.

Exclusion Criteria:

* Patients with metastatic disease, known prior to surgery.
* Patients in whom surgical resection is planned without curative intent.
* Patients who have undergone neoadjuvant treatment.
* Patients with renal failure, measured by creatinine level >1.5
* Patients with significant heart failure (NYHA functional class 3 or higher)
* Patients with significant liver failure (known cirrhosis, Bilirubin level>2)
* Patients suffering from asthma
* Patients with known allergy to one or more of the study medications
* Patients with known allergy to any medication from the non-steroidal anti-inflammatory drug group.
* Patients with diabetes mellitus (type 1 or 2).
* Patients treated chronically with one or more of the study medications
* Patients treated chronically with any type of Beta adrenergic blocker.
* Patients treated chronically with any type of COX inhibitor.
* Patients with second or third degree AV block.
* Patients with sinus bradycardia (patients with heart rate of less than 50).
* Patients with sick sinus syndrome.
* Patients with current atrial fibrillation/flutter.
* Patients with Printzmetal's angina
* Patients with hypertension
* Patients with right sided heart failure owing to pulmonary hypertension.
* Patients with significant cardiomegaly
* Patients with (current) pheochromocytoma
* Patients with chronic Digoxin treatment
* Patients with active peptic disease
* Patients with peripheral vascular disease
* Patients with history or concomitant malignant disease of any type other than breast cancer.
* Patients who were treated with chemotherapy in the last 10 years for any reason besides neo-adjuvant therapy for breast cancer within the last six months.
* Pregnant woman.
* Patients currently participating in any other clinical trial

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2014-06; Primary Completion 2016-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
No. & cytotoxic activity of NK cells, levels of NKT cells, lymphocytes, monocytes and granulocytes; cytokine levels; In vitro cytokine secretion; levels of cortisol and VEGF. Cancer recurrence in 5 years | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Tanir M Allweis, MD, Principal Investigator — Kaplan Medical Center; Shamgar Ben-Eliyahu, PhD, Study Director — Tel Aviv University, Neuroimmunology Research Unit; Moshe Shabtai, MD, Principal Investigator — Sheba Medical Center; Eran Sharon, MD, Principal Investigator — Rabin Medical Center
Locations (3):
- Israel (3):
  - Rabin Medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Kaplan Medical Center, Rehovot